CLINICAL TRIAL: NCT01705353
Title: Pilot Study of the Role of HMGB-1 in Retarding Recovery in Chronic Stroke
Brief Title: The Role of HMGB-1 in Chronic Stroke
Status: Terminated | Type: Observational
Why Stopped: study stopped because patient access became extremely limited for the initial data entry point.
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Bruce Volpe, Investigator (MD), Northwell Health
Other Study IDs: 12-090B
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Cerebrovascular Accident; Cerebral Stroke; Stroke, Acute
Keywords: Stroke; Cerebrovascular Accident; HMGB-1; cytokines; functional recovery; inflammation; immune response
MeSH Terms: conditions — Stroke; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, DNA, serum/serum cytokines
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to measure the presence of HMGB-1 and other proteins in the blood across five time points after stroke, and to determine if their presence correlates with rate of stroke recovery.

DETAILED DESCRIPTION:
Stroke, cerebrovascular accident, is the leading cause of brain injury and the leading cause of permanent disability. The acute pathophysiology of stroke depends on the innate immune response, which arises from mostly pro-inflammatory cascades. The chronic pathophysiology of stroke is less clear as the innate inflammatory response fades and matures into an adaptive immune response. HMGB-1 is a serum cytokine that has been found with persistent elevated levels for weeks to months after neurological insult in preclinical experiments, and may retard functional recovery. Elucidation of the relationship between HMGB-1 levels and the rate of functional recovery after stroke could lead to a better understanding of the systemic inflammatory response and more targeted therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the stroke service at Northshore and LIJ Medical Centers
* Patients 18 years of age or older

Exclusion Criteria:

* Patients < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute care hospital (stroke unit)
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Cytokine levels (HMGB-1) in plasma samples | day 1, day7, day 14, day 30, day 90

SECONDARY OUTCOMES:
NIH and Rankin Clinical Measures of functional recovery | day 1, day7, day 14, day 30, day 90

CONTACTS AND LOCATIONS:
Overall Officials: Bruce T Volpe, MD, Principal Investigator — Feinstein Institute for Medical Research
Locations (2):
- United States (2):
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York

REFERENCES:
- [Background] Muhammad S, Barakat W, Stoyanov S, Murikinati S, Yang H, Tracey KJ, Bendszus M, Rossetti G, Nawroth PP, Bierhaus A, Schwaninger M. The HMGB1 receptor RAGE mediates ischemic brain damage. J Neurosci. 2008 Nov 12;28(46):12023-12031. doi: 10.1523/JNEUROSCI.2435-08.2008. PMID 19005067
- [Background] Goldstein RS, Gallowitsch-Puerta M, Yang L, Rosas-Ballina M, Huston JM, Czura CJ, Lee DC, Ward MF, Bruchfeld AN, Wang H, Lesser ML, Church AL, Litroff AH, Sama AE, Tracey KJ. Elevated high-mobility group box 1 levels in patients with cerebral and myocardial ischemia. Shock. 2006 Jun;25(6):571-4. doi: 10.1097/01.shk.0000209540.99176.72. PMID 16721263

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT01705353/Prot_SAP_000.pdf